CLINICAL TRIAL: NCT02174042
Title: The Effect of Tang Ning Tongluo Formula, a Traditional Chinese Miao Medicine, in Type 2 Diabetics: A Retrospective Clinical Analysis
Brief Title: The Effect of Tang Ning Tongluo Formula in Type 2 Diabetics Clinical Analysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guizhou Bailing Group Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNTL-14-03
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: General Disorders and Administration Site Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tangning Tongluo Capsule (Experimental): Type 2 diabetes
  Interventions: Drug: Tangning Tongluo Capsule

INTERVENTIONS:
Drug: Tangning Tongluo Capsule — Taken drugs 3 times a day, with each time 3 grains
  Other Names: TNTL Capsule

SUMMARY:
The aim of this retrospective study is to review and describe safety and efficacy of Tang Ning Tong Luo capsule.

DETAILED DESCRIPTION:
The aim of this retrospective study is to review and describe safety and efficacy of Tang Ning Tong Luo capsule,a traditional Chinese Miao medicine, in Type 2 Diabetics.

ELIGIBILITY:
Inclusion criteria:

1. diagnosis of type 2 diabetes for more than one year.
2. the sustained follow-up time >3 month.
3. TNTL single or combined treatment time >3 month.
4. Chinese ethnicity.

Exclusion criteria:

1. the medical record information is not original and available.
2. lactating or pregnant.
3. diagnosis of heart failure, acute myocardial infarction, stroke, or serious injuries.
4. any other conditions not suitable for trial as evaluated by the physician in charge.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The Changing (%) of Blood Glucose Level and Glycosylated Hemoglobin Level from Baseline | At least 3 months
  The Changing (%) of Blood Glucose Level (mmol/L) and Glycosylated Hemoglobin Level (%) from Baseline (start using Tang Ning Tong Luo capsule) in recruited Type 2 diabetes patients.

SECONDARY OUTCOMES:
The Number of Participants with Adverse Events Using Tangning Tongluo Capsule | At least 3 months
  The Number of Participants with Adverse Events Using Tangning Tongluo Capsule in the Treatment ofType II Diabetes

OTHER OUTCOMES:
Number of adverse events in recruited patients. | At least 3 months
  Number of adverse events in recruited patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wenshu Teng, Dr., Study Director — ICMJE
Locations (1):
- Nanmeng Tianyuan hospital; Dongfang Hospital; China-Japanese Friendship Hospital, Beijing Shi, Guizhou, China